CLINICAL TRIAL: NCT01988207
Title: Treating Laryngeal Hyperfunction With Flow Phonation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Central Arkansas (Other)
Responsible Party: Principal Investigator, Gary H. McCullough, Professor, Interim Dean of Graduate School, University of Central Arkansas
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13-135
Record Dates: First submitted 2013-09-16; First posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Muscle Tension Dysphonia
Keywords: Muscle Tension Dysphonia; Voice; Hyperfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12 Exercise Sessions (Experimental): Patients will receive 12 treatment sessions with flow phonation exercises, as well as education on vocal hygiene.
  Interventions: Behavioral: Vocal Hygiene Training; Behavioral: Flow Phonation Exercises
- 6 Hygiene and 6 Exercise (Active Comparator): Patients will receive 6 sessions of vocal hygiene training for initial comparison to patients in Arm 1. They will then receive 6 sessions of vocal exercise training and vocal hygiene training combined.
  Interventions: Behavioral: Vocal Hygiene Training; Behavioral: Flow Phonation Exercises

INTERVENTIONS:
Behavioral: Vocal Hygiene Training — Patients will receive education on how to care for their voices on three factors: 1) hydration, 2) exogenous inflammation control, and 3) abstinence of yelling and screaming.
Behavioral: Flow Phonation Exercises — Three exercises are employed: gargling, cup bubble blowing, and stretch and flow (tissue blowing). Each is done without voicing, with voicing, and then with variations in pitch and verbalization.

SUMMARY:
The purposes of the proposed study are: a) to determine whether Flow Phonation can decrease Laryngeal Resistance (Rlaw) in patients with Muscle Tension Dysphonia (MTD); and b)establish the relationship between changes in measures of Rlaw and phonatory airflow to endoscopic, perceptual, acoustic, and handicap assessment ratings. MTD can have a debilitating effect on individuals who rely on their voices the most-teachers, preachers,salespeople, singers-costing them time, money, and even their jobs. It can lead to vocal fatigue, pain, and complete loss of voice. While treatments have emerged with some promising effects, no treatments have proven to have long-term benefits to all patients. Our preliminary data demonstrate Flow Phonation training resulted in significant decreases in Laryngeal Resistance to phonatory airflow with associated improvements in voice quality and voice handicap ratings. Sample size for our pilot study was small; no control group was utilized; and outcome measures were limited. In the proposed investigation, a larger sample will be obtained, a control group of participants receiving only Vocal Hygiene Training will be used for comparison during the first 3 weeks, and a wider range of outcome measures will be included over a longer period of time (1 year).

DETAILED DESCRIPTION:
All participants will complete the Evaluation Protocol at baseline, after 3 weeks (PERIOD 1),after 6 weeks (PERIOD 2), and for follow-up at 3, 6, and 12 months post-treatment. During PERIOD 1 (first 3 weeks), participants in ARM 1 will receive Vocal Hygiene Training as well as Airflow Exercise Training and participants in ARM 2 (the Control Arm) will receive only Vocal Hygiene Training. Vocal hygiene training alone has been demonstrated to have minimal impact on voicing32-34. During Period 2 (second 3 weeks), participants in BOTH ARMS will receive Vocal Hygiene Training and Airflow Exercise Training (Fig 3). Thus, participants in Arm 2 will receive no Flow Phonation for initial controlled comparison then 3 weeks of Flow Phonation for dose response comparison to Arm 1 (non-control) participants.

Assessment Protocol

Each participant will receive the Complete Evaluation Protocol at Baseline, after 3 weeks(PERIOD 1), after an additional 3 weeks (PERIOD 2), as well as at 3, 6, and 12 months posttreatment. These will include:

a. Laryngostroboscopic Examination b) Perceptual Voice Analysis/CAPE-V48-49 c) Acoustic Analysis/Computerized Speech Lab(CSL, KayPENTAX Corp) d) Aerodynamic Analysis/The KayPENTAX Phonatory Aerodynamic System (PAS) Model 6600 (KayPENTAX Corp.

e) Patients' Perception of Voice Handicap/Voice Handicap Index

Treatment Protocol Flow Phonation Each treatment session will take place in the same clinical room as the assessment and utilize three exercises: gargling, cup bubble blowing, and stretch and flow. Each exercise uses a built in form of biofeedback (water or tissue) and the same basic progression of activities (with minor alterations): 1) airflow task without voicing to establish positive airflow; 2) adding voicing to the task; 3) moving up and down the pitch range during the voicing task; 4) moving to a speaking/voicing task; and 5) removing biofeedback. During each vocalization attempt, the clinician listens for a clear and effortless vocal quality and trains the participant to listen.

Vocal Hygiene Training Vocal hygiene training centers on three factors: 1) hydration, 2) exogenous inflammation control, and 3) abstinence from yelling and screaming. Information will be provided initially as a Powerpoint presentation, during which each participant will have a manual and will write down answers to specific questions. Based on responses to the questions, the study clinician, in concert with the participant, will develop a set of recommendations for vocal hygiene. Examples of potential vocal hygiene targets are provided in Table 2. Three to five recommendations will be targeted for each participant, based on clinical judgment, although these numbers will serve only as a guide.

Participants will be provided a daily log to utilize where they can mark each target daily and make comments on how the target was met or not met. Each treatment session where Vocal Hygiene Training is targeted, alone or in concert with Airflow Training, participants will first present their goals, then provide the daily log and discuss successes and failures since the prior session. The study clinician and participant will then discuss the benefits of the successes and problem solve ways to improve upon failures.

ELIGIBILITY:
Inclusion Criteria:

* Rlaw greater than 1 standard deviation above or below mean
* Voice Handicap Index of greater than 18
* CAPE-V severity of 20 or greater
* willing to sign informed consent
* women must not have experienced menopause or be pregnant

Exclusion Criteria:

* organic lesion of the vocal folds
* history of neurologic disease
* history of head and neck cancer
* pulmonary disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Laryngeal Airway Resistance (Rlaw) Change Over Time | 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months
  Measured using the KayPENTAX Phonatory Aerodynamic System during a voice efficiency task (i.e., repeating "apapapapapapapa."

SECONDARY OUTCOMES:
Voice Handicap Index (VHI) | 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months
  The Voice Handicap Index is a 30 item questionnaire to assess the patient's perception of the impact of their voice on their quality of life and daily functioning.
Consensus Auditory Perceptual Evaluation - Voice | 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months
  The CAPE-V is a perceptual measure of voicing made by the clinician to rate the patient's vocal quality on a 100 mm line scale.
Noise-to-Harmonic Ratio | 3 weeks, 6 weeks, 12 weeks, 3 months, 12 months
  The KayPENTAX Computerized Speech Lab will be used to record and analyze sustained phonation (AH) and provide a measure of noise to harmonic ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Gary H McCullough, Ph.D., Principal Investigator — University of Central Arkansas
Locations (1):
- University of Central Arkansas, Conway, Arkansas, United States